CLINICAL TRIAL: NCT00692393
Title: Primary vs. Secondary Anastomosis After Sigmoid Colon Resection for Perforated Diverticulitis (Hinchey Stage III and IV): a Prospective Multicentric Randomized Trial
Brief Title: Primary vs. Secondary Anastomosis for Hinchey Stage III-IV Diverticulitis a Prospective Randomized Trial
Acronym: DIVERTI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Rouen (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2006/103/HP
Record Dates: First submitted 2008-06-03; First posted 2008-06-06 (Estimated); Last update posted 2014-06-19 (Estimated); Status verified 2014-06

CONDITIONS: Peritonitis
MeSH Terms: conditions — Peritonitis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Active Comparator): Surgery : Hartmann intervention
  Interventions: Procedure: Hartmann intervention
- 2 (Experimental): Surgery : primary resection with anastomosis with protective stoma
  Interventions: Procedure: Protected anastomosis resection

INTERVENTIONS:
Procedure: Hartmann intervention — sigmoid resection, peritoneal and rectal lavage, terminal stoma
  Arms: 1
Procedure: Protected anastomosis resection — sigmoid resection , peritoneal and rectal lavage, anastomosis, diverting stoma
  Arms: 2

SUMMARY:
This study compares primary resection with anastomosis and Hartmann's procedure in an adult population with acute perforated colonic diverticulitis (Hinchey Stage III and IV) METHODS: The primary end point was postoperative mortality. Secondary end points included surgical and medical morbidity, operative time, and length of postoperative hospitalization.

DETAILED DESCRIPTION:
inclusion criteria: hinchey III and IV diverticulitis

ELIGIBILITY:
Inclusion Criteria:

* Patient with peritonitis du to sigmoid diverticulum complication
* Surgeon - anesthetist confirming the 2 surgeries can be performed

Exclusion Criteria:

* Physical state which can not permit patient to participate
* contraindication to surgery
* non-diverticulum peritonitis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 102 (Actual)
Dates: Start 2008-06; Primary Completion 2012-12 (Actual); Study Completion 2013-11 (Actual)

PRIMARY OUTCOMES:
Death rate comparison between two chirurgical strategies | 18 months

CONTACTS AND LOCATIONS:
Overall Officials: JJ TUECH, PhD, Principal Investigator — UH Rouen
Locations (1):
- CHU - Rouen, Rouen, France